CLINICAL TRIAL: NCT00482937
Title: A Phase I, Single Ascending Dose Trial to Examine the Safety and Pharmacodynamic Effects of CD-NP
Brief Title: Safety and Pharmacodynamic Study of CD-NP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nile Therapeutics (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NIL-CDNP-CT001
Record Dates: First submitted 2007-06-04; First posted 2007-06-06 (Estimated); Last update posted 2007-06-06 (Estimated); Status verified 2007-06

CONDITIONS: Heart Failure, Congestive
Keywords: Safety; Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: CD-NP

SUMMARY:
The primary objective of this study is to establish the safety of CD-NP in normal human volunteers.

DETAILED DESCRIPTION:
The study will be conducted in two phases. The first phase, "ascending dose phase", will be an open-label study in cohorts of four (4) subjects (entered two subjects at a time) with the primary objective of establishing the safety of CD-NP. The second phase, "MTD confirmation phase", will be conducted under randomized, double-blind, placebo-controlled conditions in a larger cohort of subjects (10 subjects). The primary objective of this phase will be to confirm the safety and pharmacodynamic findings at the apparent MTD.

Secondary objectives include evaluation of the effect of CD-NP on: mean arterial pressure (MAP), heart rate (HR), urinary sodium and potassium excretion (UNaV and UKV, respectively), urinary flow rate (UV), and creatinine clearance. Plasma concentrations of CD-NP, angiotensin II, and aldosterone, and the urinary excretion rates of cGMP and CD-NP will also be determined.

ELIGIBILITY:
Inclusion Criteria:

* Be a healthy male using reliable contraception, a post-menopausal female, or a surgically sterilized female 18 to 60 years of age
* Have a BMI within the range of 18-34 kg/m2
* Be able to communicate effectively with the study personnel
* Have no significant disease or abnormal laboratory values as determined by medical history, physical examination or laboratory evaluations, conducted at the screening visit or on admission to the clinic
* Have a normal 12-lead electrocardiogram, without any clinically significant abnormalities
* Be nonsmokers defined as not having smoked in the past 6 months
* Be adequately informed of the nature and risks of the study and give written informed consent prior to receiving study medication

Exclusion Criteria:

* Known hypersensitivity or allergy to CD-NP or its components, nesiritide, other natriuretic peptides, or related compounds
* Women who are pregnant or breast-feeding
* Any disease or condition (medical or surgical) which, in the opinion of the investigator, might compromise the hematologic, cardiovascular, pulmonary, renal, gastrointestinal, hepatic, or central nervous system; or other conditions that may interfere with the absorption, distribution, metabolism or excretion of study drug, or would place the subject at increased risk
* The presence of abnormal laboratory values which are considered clinically significant.
* Positive screen for Hepatitis B (HbsAg, Hepatitis B Surface Antigen), Hepatitis C (anti HCV, Hepatitis C Antibody), or HIV (anti-HIV 1/2).
* Received an investigational drug within a period of 30 days prior to enrollment in the study.
* Received any drug therapy within 1 week, or 5 half-lives, prior to administration of the first dose of any study-related treatment. This exclusion is extended to 4 weeks for any drugs known to induce or inhibit hepatic drug metabolism. Use of NSAIDs, sulfonamides, probenecid or other drugs known to alter renal or tubular function is specifically prohibited for at least 5 half-lives prior to the first dose of any study related treatment.
* Consumption of alcohol within 48 hours prior to dose administration or during any in-patient period.
* A positive urine drug screen including ethanol, cocaine, THC, barbiturates, amphetamines, benzodiazepines, and opiates.
* A history (within the last 2 years) of alcohol abuse, illicit drug use, significant mental illness, physical dependence to any opioid, or any history of drug abuse or addiction.
* A history of difficulty with donating blood. Donated blood or blood products within 45 days prior to enrollment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2007-01; Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- DaVita Clinical Research, Minneapolis, Minnesota, United States